CLINICAL TRIAL: NCT03113279
Title: Influence of Increasing Physical Activity on Body Composition, Metabolic Health and Muscle Anabolism in Old Obese Adults
Brief Title: Mechanisms of Age-Related Muscle Loss
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: RG-13_183
Record Dates: First submitted 2017-03-28; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Sarcopenic Obesity; Muscle Weakness; Protein Metabolism Disorder; Physical Activity
MeSH Terms: conditions — Muscle Weakness; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese older individuals: Obese older individuals
- Lean older individuals: Lean older individuals
- Young lean individuals: Young lean individuals

SUMMARY:
Two independent, but interrelated conditions that have a growing impact on healthy life expectancy and health care costs in developed nations are the age related loss of muscle mass (sarcopenia) and obesity. Sarcopenia affects approximately one third of adults over 60 years of age and more than 50% of those over 80 years, which is of concern when one considers that the most rapidly expanding population demographic in the UK is adults >80 years of age.

Skeletal muscle is important in regulating blood glucose and insulin sensitivity. Thus, sarcopenia may play a role in exacerbating insulin resistance and progression toward Type II diabetes (T2D). Indeed, the highest incidence of T2D in the UK has been noted to occur in adults >65 years. Obesity is a major risk factor for chronic diseases including T2D and cardiovascular disease. Progression towards obesity is associated with a concomitant decrease in muscle mass, producing an unfavorable ratio of fat to muscle. Thus, obesity in old age may exacerbate the progression of sarcopenia.

For the proposed study the investigators will conduct preliminary laboratory tests to characterize body composition, insulin sensitivity, systemic inflammation, aerobic capacity and muscle protein metabolism (in the fasted and fed state) in healthy older and obese older adults for comparison against healthy young individuals.

DETAILED DESCRIPTION:
Twenty healthy young (aged 18-35), healthy old and obese older adults (aged ≥65) will be recruited. Old groups will be matched for age and sexual dimorphism. Obese participants will be classed as prediabetic based on a fasting A1C between 5.7 and 6.4% and impaired fasting glucose between 5.6 and 6.9 mmol/L. Obese participants will habitually take between 2000-5000 steps per day, whilst healthy young and old participants will complete >5000 steps per day.

VISIT 1 Preliminary assessments - Over a 3day period, participants will be instructed to wear a portable pedometer, to allow visual feedback on step count, and an armband accelerometer to determine habitual daily energy expenditure and the intensity of physical activity. In addition, participants will log their dietary intake.

VISIT 2 Body composition and metabolic profiling After consuming a standardized meal the previous evening, participants will report to the Wellcome Trust Clinical Research Facility in a 10 hour fasted state at approximately 09.00. Participants will be weighed in light clothing and blood pressure will be measured. Thereafter, body composition will be determined using dual energy Xray absorptiometry (DXA) and resting metabolic rate (RMR) via ventilated hood and continuous gas collection. Following RMR, a catheter will be inserted into a forearm vein and a resting, fasted blood sample obtained to determine postprandial insulin sensitivity using the HOMA-IR index.

VISIT 3 Muscle protein metabolism Participants will return to the lab in a 10 hour fasted-state at approximately 07.00 having refrained from strenuous exercise for 48 hours previously. Catheters will be inserted into the antecubital vein of both forearms. A primed, continuous infusion of isotopically labeled amino acid will be infused into one arm and the other will be used for frequent blood sampling. Muscle biopsies will be obtained 3 and 7 hours into the infusion to determine postabsorptive and postprandial rates of muscle protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 65-85 years old for older individuals and 18-35 years for younger individuals
2. Sex: Men and women
3. BMI: 18-25 kg/m2 for healthy non-obese young and elderly control group and >30 kg/m2 for obese older participants.
4. Diagnosis / General Health: For healthy elderly, good general health (no known cardiovascular or metabolic disease), nonsmokers, accustomed to normal levels of activity as assessed by pedometer and accelerometer devices during baseline testing (>5000 steps per day). For obese elderly, general good health (no known cardiovascular or metabolic disease), nonsmokers, with low levels of physical activity as assessed by pedometer and accelerometer devices during baseline testing (<4000 steps per day). Fasting blood glucose must be <5.6 mmol/mL for healthy older adults and between 5.6 and 6.9 mmol/mL for obese older adults. Fasting concentrations of A1C should be <5.7% for healthy and between 5.7 and 6.4% for prediabetic older adults. These values are in line with the type 2 diabetes classification listed by The American Diabetes Association (DIABETES CARE, VOLUME 33, SUPPLEMENT 1, JANUARY 2010).
5. Compliance: understands and is willing, able and likely to comply with all study procedures and restrictions.
6. Consent: demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent.

Exclusion Criteria:

1. Health problems such as: heart disease, rheumatoid arthritis, diabetes, poor lung function, uncontrolled hypertension, or any health conditions that might put the participant at risk for this study.
2. Recent failure to obtain clearance for exercise participation from family physician/medical doctor.
3. Regular consumption of any analgesic or anti-inflammatory drug(s), prescription or nonprescription.
4. Taking any medications known to affect protein metabolism (i.e. b-blockers, corticosteroids, nonsteroidal anti-inflammatories, or prescription strength acne medications). Medications will be deemed inappropriate based on the Chief Investigators discretion
5. Individuals who complete fewer than 1000 steps per day (as assessed by pedometer prior to the study) or those who participate in regular structured exercise (running or strength training) more than 2 times per week.
6. Participants will be excluded if they fail to comply with the physical activity demands of the study. Exclusion will occur if the following are not met. Failure to meet the expected daily step count target on more than one occasion per week during the 21 day intervention will be deemed as failure to comply.
7. Participants who have previously (within 5 years of the present study) undergone infusion of an amino acid tracer and/or had 4 or more muscle biopsies obtained from the quadriceps region will be excluded.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: * Young lean healthy inidivduals aged 18-35.
  * Lean healthy older individuals aged 65-85.
  * Obese inactive older individuals aged 65-85.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein synthesis rates via mass spectrometry | 2 years
  Postabsorptive and postprandial myofibrillar protein synthesis rates between groups and following the activity intervention

SECONDARY OUTCOMES:
Muscle fibre properties via immunohistochemical staining | 2 years
  muscle fibre type (i.e. I and II) and cross sectional area
Muscle fibre lipid content immunofluorescent staining | 2 years
  Intramyocellular lipid content in Type I and II fibres
Physical activity levels via accelerometry | 2 years
  Daily average time spent in sedentary, light, moderate or vigorous intensity activity
Inflammation via plasma/insulin assays | 2 years
  Blood markers of inflammation, interleukin 6 and c-reactive protein
Insulin sensitivity via plasma assays | 2 years
  Blood samples will be analyzed for insulin, glucose and hbA1C for indication of whole-body insulin sensitivity
Body composition via dual x-ray absorptiometry | 2 years
  DXA-derived fat and fat free mass will be measured
Intramuscular signaling via western blot | 2 years
  Western blots for phosphorylation of key anabolic signaling proteins
Dietary intake via dietary logs | 2 years
  Diet logs will be assessed for total energy and macronutrient intake
Daily step count by pedometer | 2 years
  Average daily step count assessed via waist worn pedometer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smeuninx B, Mckendry J, Wilson D, Martin U, Breen L. Age-Related Anabolic Resistance of Myofibrillar Protein Synthesis Is Exacerbated in Obese Inactive Individuals. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3535-3545. doi: 10.1210/jc.2017-00869. PMID 28911148